CLINICAL TRIAL: NCT05559047
Title: Field Usability Study of Eclipse CPAP Device
Brief Title: Field Usability Study of Eclipse Mask
Status: Completed | Type: Observational
Sponsor: Bleep, LLC (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: BSL-SNAP-002; 1R44HL158286-01A1 (NIH)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- In-House Usability Study Group: Seventy adherent CPAP users will volunteer to trial the Eclipse mask for two nights in their homes. Participants who attend an appointment at one of three offices of Sleep Centers of Middle Tennessee (SCMT) and will be trained how to use the Eclipse mask, then asked to use the Eclipse for two consecutive nights and then complete a participant survey after the second night.
  Participants will follow instructions to set up and put on the Eclipse nasal mask.
  They will fill out a survey about the ease and comfort of putting on and wearing the mask, briefly.
  Interventions: Device: Eclipse mask

INTERVENTIONS:
Device: Eclipse mask — Users will interact with the Eclipse CPAP machine and report on usability/likeability.

SUMMARY:
The study is designed to assess the usability of a novel CPAP human interface compared to a traditional nasal mask. Human subjects will interact with two different CPAP interfaces including a traditional CPAP mask and the 2nd generation DreamPort-Eclipse. Subjects will be requested to put on each of the different CPAP interface options a total of three times for a total of 6 trials. The order of device will be randomized.

ELIGIBILITY:
Inclusion Criteria:

•Male or female ≥18 years old who are impacted by obstructive sleep apnea and currently are familiar with a CPAP device.

Exclusion Criteria:

* Diagnosis of any medical or behavioral conditions that would compromise subject safety.
* Under the age of 18: target for this current version of the platform is the adult population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults over the age of 18 who are CPAP users and attend SCAT centers who volunteer to be in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Heatherington, Principal Investigator — Bleep, LLC
Locations (3):
- United States (3):
  - AeroFlow Sleep, Asheville, North Carolina
  - Advanced Respiratory and Sleep Medicine, Huntersville, North Carolina
  - Sleep Centers of Middle Tennessee, Murfreesboro, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Data collected through surveys will be available upon request to the principal investigator. Data requested will be de-identified. Only de-identified data will be made available. Only survey responses and the investigators' observational notes, also deidentified, will be shared. No PHI will be shared. Aggregated participant demographic data will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available 4 years after the study completion.
Access Criteria: Requests will be made in writing, to the PI, at stuart@bleepsleep.com. Requests should include the reason for the request, how the data is intended to be used, and additional information may be requested. Data will be shared with credentialed, licensed, or otherwise verifiable researchers/investigators for research purposes only.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, seventy adherent CPAP users volunteered to trial the Eclipse mask for two nights in their homes. Participants attended an appointment at one of three offices of Sleep Centers of Middle Tennessee (SCMT) and were trained how to use the Eclipse mask, then asked to use the Eclipse for two consecutive nights and then complete a participant survey after the second night. No control group was used. Volunteers were gathered from the pool of SCMT participants.
Groups:
- Eclipse Mask Group (Single Arm Study): A single group was used, namely those trying the Eclipse mask at home for 2 nights
Period: Overall Study
Arm/Group | Eclipse Mask Group (Single Arm Study)
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Seventy adherent CPAP users volunteered to trial the Eclipse mask for two nights in their homes. Participants attended an appointment at one of three offices of Sleep Centers of Middle Tennessee (SCMT) and were trained how to use the Eclipse mask, then asked to use the Eclipse for two consecutive nights and then complete a participant survey after the second night. The volunteers were selected to cover a demographic range of races and gender as required by study sponsor.
Groups:
- Eclipse Mask (Single Arm Study): Seventy adherent CPAP users will volunteer to trial the Eclipse mask for two nights in their homes. Participants who attend an appointment at one of three offices of Sleep Centers of Middle Tennessee (SCMT) and will be trained on how to use the Eclipse mask, then asked to use the Eclipse for two consecutive nights and then complete a participant survey after the second night.
  Eclipse novel CPAP mask: Participants will follow instructions to set up and put on the Eclipse nasal mask. The Eclipse removes the headgear associated with traditional CPAP masks, offering a small compact design weighing less than an ounce. The Eclipse uses small and lightweight adhesive seals around the nostrils to create an ergonomic design which accommodates the shape of each individual user. It completes a perfect circuit for CPAP therapy to deliver pressure to the airway and stabilize the user's disordered breathing during sleep (apnea and snoring).
  Participants will follow instructions to set up and put on the mask. They will fill out a survey about the ease and comfort of putting on and wearing the mask, briefly.
Arm/Group | Eclipse Mask (Single Arm Study)
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants] — Participant must be 18 years or older.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 68
    >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 44
Race/Ethnicity, Customized [Number; unit: participants]
  White | 23
  Black | 26
  Hispanic | 14
  Asian | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Asked for Additional Information
Description: The total count of participants who asked for additional information during the course of home use of the mask was recorded
Time Frame: Throughout the duration of the study (48 hours)
Measure: Count of Participants; unit: Participants
Groups:
- Eclipse Novel CPAP Mask: Participants will follow instructions to set up and put on the Eclipse nasal mask. The Eclipse removes the headgear associated with traditional CPAP masks, offering a small compact design weighing less than an ounce. The Eclipse uses small and lightweight adhesive seals around the nostrils to create an ergonomic design which accommodates the shape of each individual user. It completes a perfect circuit for CPAP therapy to deliver pressure to the airway and stabilize the user's disordered breathing during sleep (apnea and snoring).
Arm/Group | Eclipse Novel CPAP Mask
Number analyzed (Participants) | 70
Participants | 6

2. Primary Outcome: Mask Likeability
Description: A 16-item patient survey was administered to the participants at the end of the study. Patients had to answer according to a Likert scale (1: worst, 5:best). Here, this reflects the average of all the answered items. For example, question number one had an average score of 4.52, question number 2 had an average score of 4.21, etc. Since all questions reflect mask likability, they were averaged to provide an overall score.
Time Frame: At 48 hours
Measure: Mean (Standard Deviation); unit: score
Groups:
- Eclipse Novel CPAP Mask: Participants will follow instructions to set up and put on the Eclipse nasal mask. The Eclipse removes the headgear associated with traditional CPAP masks, offering a small compact design weighing less than an ounce. The Eclipse uses small and lightweight adhesive seals around the nostrils to create an ergonomic design which accommodates the shape of each individual user. It completes a perfect circuit for CPAP therapy to deliver pressure to the airway and stabilize the user's disordered breathing during sleep (apnea and snoring).
  Participants will follow instructions to set up and put on the mask. They will fill out a survey about the ease and comfort of putting on and wearing the mask, briefly.
Arm/Group | Eclipse Novel CPAP Mask
Number analyzed (Participants) | 70
score | 4.1 (0.4)

3. Primary Outcome: Number of Participants Who Experienced Technical Issues
Description: Total count of participants who reported technical issues during the course of the 48 h home use of the mask were recorded
Time Frame: The duration of the trial (48 h)
Measure: Count of Participants; unit: Participants
Arm/Group | Eclipse Novel CPAP Mask
Number analyzed (Participants) | 70
Participants | 7

ADVERSE EVENTS:
Time Frame: Participants wore the mask for a 2 night duration and occurrence of adverse events was assessed throughout this time
Groups:
- Eclipse Novel CPAP Mask: Seventy adherent CPAP users will trial the Eclipse mask for two nights in their homes. Participants who attend an appointment at one of three offices of Sleep Centers of Middle Tennessee (SCMT) and will be trained on how to use the Eclipse mask, then asked to use the Eclipse for two consecutive nights and then complete a participant survey after the second night. No control group was used.
  Eclipse novel CPAP mask: Participants will follow instructions to set up and put on the Eclipse nasal mask. The Eclipse removes the headgear associated with traditional CPAP masks, offering a small compact design weighing less than an ounce. The Eclipse uses small and lightweight adhesive seals around the nostrils to create an ergonomic design which accommodates the shape of each individual user. It completes a perfect circuit for CPAP therapy to deliver pressure to the airway and stabilize the user's disordered breathing during sleep (apnea and snoring).
  Participants will follow instructions to set up and put on the mask. They will fill out a survey about the ease and comfort of putting on and wearing the mask, briefly.
Arm/Group | Eclipse Novel CPAP Mask
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT05559047/Prot_SAP_000.pdf